CLINICAL TRIAL: NCT02753036
Title: Chemotherapy-induced Cognitive Alterations in Recruits With Ovarian and Breast Cancer (CICARO)
Brief Title: Chemotherapy-induced Cognitive Alterations in Recruits With Ovarian and Breast Cancer
Acronym: CICARO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Petra Huehnchen, resident and postdoctoral fellow, Charite University, Berlin, Germany
Other Study IDs: EA4/069/14
Record Dates: First submitted 2016-04-20; First posted 2016-04-27 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Cognition Disorders; Polyneuropathies
Keywords: cognition; chemotherapy; polyneuropathy; paclitaxel; cancer; chemobrain
MeSH Terms: conditions — Cognition Disorders; Polyneuropathies; Neoplasms; Chemotherapy-Related Cognitive Impairment | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum samples, PBMC
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Chemotherapy: patients with ovarian cancer and paclitaxel + carboplatin combination chemotherapy as well as patients with breast cancer and paclitaxel +/- carboplatin combination chemotherapy
  Interventions: Drug: Chemotherapy
- Healthy control: patients with benign gynecological tumors after laparoscopic surgical resection
- Tumor control: patients with breast cancer with anti-hormonal and/or localized radiation treatment but no chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — standard combination chemotherapy (paclitaxel +/- carboplatin) if necessary according to treatment guidelines
  Groups: Chemotherapy

SUMMARY:
Neurotoxic phenomena are among the most common and difficult to treat side effects of chemotherapy. The development of chemotherapy induced peripheral neuropathy (CIPN) is a well-recognized adverse reaction in the peripheral nervous system. Side effects of chemotherapy in the central nervous system, however, particularly changes of cognitive function (in non-medical literature referred to as "chemobrain") are diffuse and difficult to attribute to individual cytostatic drugs. The primary purpose of this study is to assess cognitive function in patients with ovarian and breast cancer before and after systemic chemotherapy with paclitaxel with standardized neuropsychological tests and compare the outcome to patients with benign gynecological tumors and breast cancer without chemotherapy treatment, respectively. Secondary parameters include the assessment of olfactory function, total neuropathy score and cytokine profiles.

DETAILED DESCRIPTION:
Primary outcome parameter:

compound score of standardized neuropsychological test

Secondary parameters:

* olfactory function (Sniffin Sticks)
* total neuropathy score (TNS), reduced version (clinical examination, neurography of sural and peroneal nerve)
* cytokine profiling from serum samples (ELISA)
* quality of life (questionnaire)
* depression screening (questionnaire)
* symptoms of polyneuropathy (questionnaire)
* symptoms of cognitive impairment (everyday memory test questionnaire)

Assessment time points:

* baseline (after surgical tumor resection and before chemotherapy)
* follow up 1 (3 weeks after last chemotherapy cycle or 21 weeks (control patients))
* follow up 2 (optional; 1 year after chemotherapy completion)

ELIGIBILITY:
Inclusion Criteria:

* age
* written informed consent
* Karnofsky index >70% / ECOG <1
* at least 8 years of education

Exclusion Criteria:

* post surgical delirium
* major depression
* alcohol or drug abuse
* anemia < 8 g/dl
* mild cognitive impairment or dementia
* previous neurotoxic chemotherapy treatment

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic, department of gynecology
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline compound score of standardized neuropsychological test | 3 weeks after last chemotherapy cycle (21 weeks)
  standardized neuropsychological test covering verbal memory, visual-spatial memory, short term/ working memory, executive functions

SECONDARY OUTCOMES:
Change from baseline olfactory function | 3 weeks after last chemotherapy cycle (21 weeks)
  standardized test battery (Sniffin Sticks)
Change from baseline total neuropathy score (TNSr) | 3 weeks after last chemotherapy cycle (21 weeks)
  reduced version includes clinical examination and neurography of sural and peroneal nerve
Change from baseline cytokine profiling (serum sample) | 3 weeks after last chemotherapy cycle (21 weeks)
  ELISA of serum samples
Change from baseline quality of life questionnaire | 3 weeks after last chemotherapy cycle (21 weeks)
  EORTC-QLQ-C30
Change from baseline depression screening questionnaire | 3 weeks after last chemotherapy cycle (21 weeks)
  DESC-I
Change from baseline symptoms of polyneuropathy questionnaire | 3 weeks after last chemotherapy cycle (21 weeks)
  EORTC-QLQ-C30+CIPN20
Change from baseline symptoms of cognitive decline (questionnaire) | 3 weeks after last chemotherapy cycle (21 weeks)
  everyday memory test

CONTACTS AND LOCATIONS:
Overall Officials: Petra Huehnchen, Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huehnchen P, Schinke C, Bangemann N, Dordevic AD, Kern J, Maierhof SK, Hew L, Nolte L, Kortvelyessy P, Gopfert JC, Ruprecht K, Somps CJ, Blohmer JU, Sehouli J, Endres M, Boehmerle W. Neurofilament proteins as a potential biomarker in chemotherapy-induced polyneuropathy. JCI Insight. 2022 Mar 22;7(6):e154395. doi: 10.1172/jci.insight.154395. PMID 35133982